CLINICAL TRIAL: NCT07343609
Title: Predictive Value of Seizure Frequency at Onset for Long-Term Seizure Control
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Farag Okaily, Postgraduate Researcher, Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: Amira Farag
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Newly Diagnosed Epilepsy With Focus on Seizure Frequency at Onset and Long-term Seizure Control
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

INTERVENTIONS:
Other: observational study (no intervention) — No intervention was applied. This is an observational study in which participants underwent routine clinical and radiological assessments only, with no experimental or therapeutic intervention.

SUMMARY:
Epilepsy is a chronic neurological disorder characterized by recurrent unprovoked seizures, and achieving long-term seizure control remains a major therapeutic goal. Early clinical features at diagnosis, particularly seizure frequency at onset and early response to antiseizure drugs (AEDs), may provide important prognostic information. Previous studies suggest that higher early seizure burden and poor initial response to AEDs are associated with unfavorable long-term outcomes; however, the predictive value of seizure frequency and number at onset remains insufficiently explored in contemporary cohorts.

This retrospective cohort study will be conducted at the Neurology Clinic of Assiut University Children's Hospital between February 2026 and January 2027. It will include patients with tractable and intractable newly diagnosed epilepsy. Data will be collected from clinical records and structured interviews, covering demographic characteristics, detailed seizure history (with emphasis on seizure frequency at onset), treatment details, early and long-term seizure control, adherence, and adverse effects. Neurological examination findings, EEG results, and neuroimaging data will be reviewed to support epilepsy classification and identify potential prognostic factors.

The primary outcome is to assess whether higher seizure frequency at onset is associated with poorer long-term seizure control. Statistical analysis will include descriptive statistics, comparative analyses between seizure-frequency groups, multivariate logistic regression to identify independent predictors, and ROC curve analysis to evaluate predictive accuracy. Ethical approval, informed consent, and data confidentiality will be ensured throughout the study.

ELIGIBILITY:
Inclusion Criteria:

- All patients with tractable and intractable epilepsy.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with tractable and intractable epilepsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
To assess whether higher seizure frequency at onset is associated with poorer long-term seizure control. | 12 months

IPD SHARING:
Plan to Share IPD: No